CLINICAL TRIAL: NCT02615314
Title: Clinical Aspects of Patients With Benign Paroxysmal Positional Vertigo (BPPV) and Migraine
Status: Completed | Type: Observational
Sponsor: Anadolu Medical Center (Other)
Responsible Party: Principal Investigator, Sertac Yetiser, Clinical Professor, Dept of ORL & HNS, Anadolu Medical Center
Other Study IDs: AnadoluMC
Record Dates: First submitted 2015-11-14; First posted 2015-11-26 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Migraine; Positional Vertigo
Keywords: migraine; benign paroxysmal positional vertigo
MeSH Terms: conditions — Migraine Disorders; Vertigo; Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- BPPV without migraine: Two hundred and sixty-three patients with BPPV (2009-2014), confirmed by videonystagmography (VNG), were enrolled in the study. Patients' charts were reviewed. They were grouped as those with or without migraine. Distribution of gender, age, duration of symptoms and affected side were reviewed. Two hundred and thirty-one patients with no migraine were identified.
  Interventions: Procedure: Particle re-positioning maneuver
- BPPV with migraine: Thirty-two patients (11.4%) with migraine were identified. Diagnosis and classification of migraine and its differentiation from other type of headaches was based on third edition of International classification of headache disorders (ICHD-III beta) by international headache society (IHS). All patients with migraine had migrainous headache with or without aura and they all were diagnosed in our institution and followed by our neurology staff.
  Interventions: Procedure: Particle re-positioning maneuver

INTERVENTIONS:
Procedure: Particle re-positioning maneuver — Patients with posterior canal BPPV (PC-BPPV) were treated with Epley maneuver. Patients with superior canal (SC-BPPV) were treated with Li or reverse Epley maneuver. Patients with lateral canal (LC) apogeotropic or geotropic nystagmus were treated with Barbeque, Semont's or Gufoni maneuvers. If geotropic or ageotropic type nystagmus is equal intensity on both sides. The involved side was determined according to the patient sense of disturbance or lying down positioning test. If the patient has involvement of both sides according to Dix-Hallpike maneuver. Therapeutic maneuver was applied to the more severe side. All patients were re-evaluated at maximum 7 days.

SUMMARY:
The aim of this study is to analyze the clinical aspects of patients with BPPV associated with migraine. It is our purpose to clarify weather migraine is a risk factor for BPPV if the clinical aspect and the therapeutic outcome is different.

DETAILED DESCRIPTION:
Two hundred and sixty-three patients with BPPV were enrolled in this retrospective study. All patients' charts were reviewed by independent observer. The type of BPPV and associated problems were noted. Patients with migraine were investigated in terms of age, gender, symptoms, affected side and the cure rate. Their data were compared with those having no migraine. Mean values and standard deviations (± SD) were calculated. One way ANOVA test was used for the analysis. Significance was set at p < 0.005.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had history of head-induced positional and brief vertigo and who have been confirmed by VNG were included

Exclusion Criteria:

* Patients with balance problem other than BPPV,
* Patients receiving any medication prior to therapeutic maneuver were excluded

Ages: 10 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: BPPV patients only confirmed by VNG
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of patients who had normal vestibular response to provocative tests 7 days after re-positioning maneuver | 7 days
  Every patient with BPPV who had positional nystagmus during Dix-Hallpike and head-roll provocative maneuvers will be treated with Epley or barbeque particle re-positioning maneuvers. Balance (positional nystagmus) of patients 7 days after re-positioning maneuvers will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Hale Gokmen, MD, Principal Investigator — Dept of Neurology, Anadolu Medical Center

REFERENCES:
- [Result] Uneri A. Migraine and benign paroxysmal positional vertigo: an outcome study of 476 patients. Ear Nose Throat J. 2004 Dec;83(12):814-5. PMID 15724736
- [Result] Ishiyama A, Jacobson KM, Baloh RW. Migraine and benign positional vertigo. Ann Otol Rhinol Laryngol. 2000 Apr;109(4):377-80. doi: 10.1177/000348940010900407. PMID 10778892
- [Result] Yetiser S, Ince D. Demographic analysis of benign paroxysmal positional vertigo as a common public health problem. Ann Med Health Sci Res. 2015 Jan-Feb;5(1):50-3. doi: 10.4103/2141-9248.149788. PMID 25745577
- [Result] von Brevern M, Radtke A, Lezius F, Feldmann M, Ziese T, Lempert T, Neuhauser H. Epidemiology of benign paroxysmal positional vertigo: a population based study. J Neurol Neurosurg Psychiatry. 2007 Jul;78(7):710-5. doi: 10.1136/jnnp.2006.100420. Epub 2006 Nov 29. PMID 17135456